CLINICAL TRIAL: NCT00514527
Title: Nuvocid® (Oritavancin) at Single or Infrequent Doses for the Treatment of Complicated Skin and Skin Structure Infections (SIMPLIFI)
Brief Title: A Study for Patients With Complicated Skin and Skin Structure Infections
Acronym: SIMPLIFI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targanta Therapeutics Corporation (Industry)
Responsible Party: Targanta Therapeutics Corporation, Targanta Therapeutics Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAR-ORI-SD001
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Staphylococcal Skin Infections; Wounds and Injuries; Abscess; Cellulitis; Streptococcal Infections
MeSH Terms: conditions — Staphylococcal Skin Infections; Wounds and Injuries; Abscess; Cellulitis; Streptococcal Infections | interventions — oritavancin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: oritavancin
- 2 (Experimental)
  Interventions: Drug: oritavancin
- 3 (Experimental)
  Interventions: Drug: oritavancin

INTERVENTIONS:
Drug: oritavancin — Oritavancin as a single, infrequent or daily dose.

SUMMARY:
Two Phase III trials to demonstrate the efficacy and safety of oritavancin in the treatment of complicated skin and skin structure infections (cSSSI) have been completed.

The pharmacokinetic profile of oritavancin in humans suggests that oritavancin has the potential to be used safely and effectively when given either as a single dose or as an infrequent dose for cSSSI. Data from animals support this theory.

SIMPLIFI has been designed to evaluate the efficacy and safety of either a single dose of oritavancin or an infrequent dose of oritavancin (First dose on Day one with an option for a second dose on Day five) compared to the previously studied dosing regimen of 200mg oritavancin given once daily for 3 to 7 days.

ELIGIBILITY:
Inclusion Criteria

* Complicated skin and skin structure infection, presumed or proven to be caused by gram-positive pathogen(s).
* Patients, ages 18 years and older, must not be below normal body weight or morbidly obese.
* Female patients must not be pregnant at time of enrollment and must agree to a reliable method of birth control during the study and for 6 months following the last dose of study drug.

Exclusion Criteria:

Patients:

* with a condition which would prevent performing protocol safety and efficacy assessments.
* who have received antibiotics for more than 24 hours within the last 3 days.
* with an infection involving deep tissues or unlikely to be caused by gram positive bacteria
* who are nursing and will not stop nursing for at least 6 months
* with a prior allergic reaction to glycopeptides (e.g. vancomycin)
* with any of the following:

  1. toxic shock syndrome or toxic-like syndrome
  2. presumed or proven infection caused by Clostridium species
  3. bone infections
  4. ischemic or gangrenous ulcers or wounds
  5. infections caused only by gram-negative bacteria
  6. infection of an artificial joint that cannot be removed
  7. infection of the scrotum, perineum or perianal region
  8. infection of a severe burn wound
  9. severe ear infection involving bone and/or cartilage
  10. infection following injury in water possibly containing Vibrio species or following a history of eating raw oysters within 1 week prior to disease onset

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Clinical success at follow-up | six months

SECONDARY OUTCOMES:
To evaluate safety of dosing regimens. | six months

CONTACTS AND LOCATIONS:
Overall Officials: Targanta Therapeutics, Study Director — simplifi@covance.com
Locations (60):
- United States (32):
  - Targanta Recruiting Site, Mobile, Alabama
  - Targanta Recruiting Site, Anaheim, California
  - Targanta Recruiting Site, Buena Park, California
  - Targanta Recruiting Site, Chula Vista, California
  - Targanta Recruiting Site, Hawaiian Gardens, California
  - Targanta Recruiting Site, Long Beach, California
  - Targanta Recruiting Site, Los Angeles, California
  - Targanta Recruiting Site, Oceanside, California
  - Targanta Recruiting Site, Rolling Hills Estates, California
  - Targanta Recruiting Site, San Jose, California
  - Targanta Recruiting Site, Torrance, California
  - Targanta Recruiting Site, Atlantis, Florida
  - Targanta Recruiting Site, Inverness, Florida
  - Targanta Recruiting Site, Miami, Florida
  - Targanta Recruiting Site, Columbus, Georgia
  - Targanta Recruiting Site, Marietta, Georgia
  - Targanta Recruiting Site, Savannah, Georgia
  - Targanta Recruiting Site, Springfield, Illinois
  - Targanta Recruiting Site, Indianapolis, Indiana
  - Targanta Recruiting Site, Baton Rouge, Louisiana
  - Targanta Recruiting Site, Lafayette, Louisiana
  - Targanta Recruiting Site, New Orleans, Louisiana
  - Targanta Recruiting Site, Cumberland, Maryland
  - Targanta Recruiting Site, Detroit, Michigan
  - Targanta Recruiting Site, Minneapolis, Minnesota
  - Targanta Recruiting Site, Albany, New York
  - Targanta Recruiting Site, Columbus, Ohio
  - Targanta Recruiting Site, Toledo, Ohio
  - Targanta Recruiting Site, Jackson, Tennessee
  - Targanta Recruiting Site, Arlington, Texas
  - Targanta Recruiting Site, Houston, Texas
  - Targanta Recruiting Site, Salt Lake City, Utah
- Australia (6):
  - Targanta Recruiting Site, Cairns, Queensland
  - Targanta Recruiting Site, Nambour, Queensland
  - Targanta Recruiting Site, Woolloongabba, Queensland
  - Targanta Recruiting Site, East Ringwood, Victoria
  - Targanta Recruiting Site, Parkville, Victoria
  - Targanta Recruiting Site, Fremantle
- India (8):
  - Targanta Recruiting Site, Hyderabaad, Andhra Pradesh
  - Targanta Recruiting Site, Ahmedabad, Gujarat
  - Targanta Recruiting Site, Vadodara, Gujarat
  - Targanta Recruiting Site, Bangalore, Karnataka
  - Targanta Recruiting Site, Kochi, Kerala
  - Targanta Recruiting Site, Mumbai, Maharashtra
  - Targanta Recruiting Site, Pune, Maharashtra
  - Targanta Recruiting Site, Lucknow, Uttar Pradesh
- Italy (6):
  - Targanta Recruiting Site, Catania
  - Targanta Recruiting Site, Mantova
  - Targanta Recruiting Site, Milan
  - Targanta Recruiting Site, Pisa
  - Targanta Recruiting Site, Savona
  - Targanta Recruiting Site, Siena
- Romania (2):
  - Targanta Recruiting Site, Bucharest
  - Targanta Recruiting Site, Craiova
- Ukraine (6):
  - Targanta Recruiting Site, Ivano-Frankivsk
  - Targanta Recruiting Site, Kharkiv
  - Targanta Recruiting Site, Kiev
  - Targanta Recruiting Site, Odesa
  - Targanta Recruiting Site, Ternopil
  - Targanta Recruiting Site, Zaporizhzhya

REFERENCES:
- [Derived] Dunbar LM, Milata J, McClure T, Wasilewski MM; SIMPLIFI Study Team. Comparison of the efficacy and safety of oritavancin front-loaded dosing regimens to daily dosing: an analysis of the SIMPLIFI trial. Antimicrob Agents Chemother. 2011 Jul;55(7):3476-84. doi: 10.1128/AAC.00029-11. Epub 2011 May 2. PMID 21537018